CLINICAL TRIAL: NCT02253225
Title: An fMRI Study of Self Processing and Self Focus in Major Depression and Bipolar Disorder
Brief Title: Self Focus in Bipolar Disorder: A Functional Magnetic Resonance Imaging (fMRI) Study
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Sharmin Ghaznavi, Staff Psychiatrist, Massachusetts General Hospital
Other Study IDs: 2012P000714; 19531 (Other Grant/Funding Number: Brain and Behavior Research Foundation)
Record Dates: First submitted 2014-09-24; First posted 2014-10-01 (Estimated); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Bipolar Disorder; Major Depression; Rumination
Keywords: Bipolar Disorder; Major Depression; Rumination; Self Processing
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Major; Rumination Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Bipolar Disorder: Clinical status will be determined using the Mini International Neuropsychiatric Interview (M.I.N.I) for 20 patients with bipolar disorder (BPAD).
  Interventions: Other: Functional Magnetic Resonance Imaging (fMRI)
- Major Depressive Disorder: Clinical status will be determined using the Mini International Neuropsychiatric Interview (M.I.N.I) for 20 patients with major depression (MDD).
  Interventions: Other: Functional Magnetic Resonance Imaging (fMRI)
- Healthy Control: Clinical status will be determined using the Mini International Neuropsychiatric Interview (M.I.N.I) for 20 normal, healthy volunteers.
  Interventions: Other: Functional Magnetic Resonance Imaging (fMRI)

INTERVENTIONS:
Other: Functional Magnetic Resonance Imaging (fMRI) — Imaging will be performed on a 3T Siemens Trio scanner. Each MRI scanning session will last no more than 90 minutes.

SUMMARY:
The investigators propose to examine both resting state activity and functional activity during rumination and during self-processing to study the relationship between neural correlates of rumination/self-focus and self-processing in major depression and bipolar disorder.

DETAILED DESCRIPTION:
Negative rumination, a specific form of self-focus, characterized by repetitively focusing on one's symptoms of distress, and the possible causes and consequences of these symptoms, is a hallmark of depression. Nearly a decade of research has culminated in evidence that the tendency to engage in negative rumination is highly correlated with depressive symptoms. Rumination also plays a critical role in the etiology and maintenance of depressed states and predicts risk for mania in bipolar disorder. Despite the central role of rumination in major depression and bipolar disorder, there have been few studies to date investigating the functional neuroanatomy of negative rumination, and no studies of positive rumination. The few neuroimaging studies that have utilized measures of the tendency to engage in negative rumination have focused on brain functioning when performing tasks that involve processing emotional or self-referential stimuli, but they have not studied resting state activity or functional activity during negative and positive rumination. We are examining both resting state activity and functional activity during negative and positive rumination and during self-processing to study the relationship between the neural correlates of rumination/self-focus and self-processing in major depression and bipolar disorder.

ELIGIBILITY:
Inclusion Criteria Healthy Controls:

* Right-handed (as determined by the Handedness Inventory; Oldfield, 1971)
* Normal or corrected-to normal vision and hearing

Exclusion Criteria for Healthy Controls:

* Any current or past psychiatric history
* Significant medical, psychiatric or neurological illness
* Currently taking antidepressants, mood stabilizers, or benzodiazepines
* Positive MR screen (e.g., metal implant, claustrophobia, etc)

Inclusion Criteria for Patients with Major Depression:

* Current diagnosis of MDD
* Right-handed (as determined by the Handedness Inventory; Oldfield, 1971)
* Normal or corrected-to normal vision and hearing

Exclusion Criteria for MDD Patients:

* If a history of substance abuse, at least 6 months in remission
* Current suicidal ideation or history of suicide attempts
* Positive MR screen (e.g., metal implant, claustrophobia, etc)

Inclusion Criteria for patients with BPAD:

* Current diagnosis of BPAD
* Right-handed (as determined by the Handedness Inventory; Oldfield, 1971)
* Normal or corrected-to normal vision and hearing

Exclusion Criteria for BPAD Patients:

* If a history of substance abuse, at least 6 months in remission
* Current suicidal ideation or history of suicide attempts
* Positive MR screen (e.g., metal implant, claustrophobia, etc)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy controls will be recruited through email announcements at MGH, internet website at Harvard, and flyers posted at the Massachusetts General Hospital and in the community (e.g., community centers, public libraries, coffee shops, restaurants, and laundromats). Subjects with major depression will be recruited through the Depression Clinic and Research Program at MGH and flyers posted at MGH. Subjects with bipolar disorder will be recruited through the Bipolar Clinic and Research Program at MGH and flyers posted at MGH.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2013-01; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Functional Magnetic Resonance Imaging (fMRI) to examine self processing and self focus | Participants will be analyzed as quickly as possible after a screening visit, an expected average of 2 weeks
  Functional Magnetic Resonance Imaging (fMRI) will be used to look at the neuroanatomy of self processing and self focus.

CONTACTS AND LOCATIONS:
Overall Officials: Sharmin Ghaznavi, M.D., Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States